CLINICAL TRIAL: NCT01910038
Title: Evaluation of Tocilizumab as an add-on Therapy to Corticoids in Giant Cell Arteritis: Proof of Concept Study.
Acronym: HORTOCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bonnotte PHRC N 2012
Record Dates: First submitted 2013-07-17; First posted 2013-07-29 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

ARMS (1):
- Prednisone+Tocilizumab (Experimental): Prednisone (0.7 mg/Kg/d and then progressively tapered to reach 0.1 mg/Kg/d at W24) + tocilizumab 8mg/Kg/4 weeks for a total of 4 infusions (S0, S4, S8, S12).
  Interventions: Drug: corticoids+ tocilizumab 8mg/Kg/4 weeks

INTERVENTIONS:
Drug: corticoids+ tocilizumab 8mg/Kg/4 weeks

SUMMARY:
It has been reported that around 40% of GCA patients are able to decrease the prednisone dose until 0.1 mg/Kg/d or less after 6 months of treatment. In this study, we hypothesized that adding 3 months of tocilizumab to prednisone could increase the percentage from 40 to 70%.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* GCA fulfilling ≥3/5 ACR criteria
* Newly diagnosed GCA or relapsing GCA if treatments (Glucocorticoids±immunosuppressants) have been stopped for at least 6 months
* Glucocorticoids started for less than 21 days
* Proof of large vessel vasculitis:

  * Positive temporal artery biopsy (TAB)
  * Aortitis, as defined by regular circumferential wall thickening ≥3mm in the absence of calcification and/or significant atheroma on angio-CT images; or a homogeneous vascular signal more intense than the liver on 18FDG-PET images.
* For men and women of a child-bearing age, an effective method of contraception must be used by the patient or his or her partner throughout the treatment with tocilizumab (or placebo) and for 3 months after the end of the treatment. Breast-feeding is not authorised until 3 months after the end of treatment with tocilizumab. Women not considered at risk of pregnancy are those defined by menopause of at least one year or surgically steriles (ligature of the fallopian tubes, bilateral ovariectomy or hysterectomy)
* Persons who have provided written informed consent
* Persons covered by the National Health Insurance Agency

Exclusion Criteria:

* Pregnancy
* hospitalization in the previous year for drug or alcohol intoxication
* current treatment for another autoimmune or inflammatory disease
* known hypersensitivity to TCZ or one of its excipients or another human or murine monoclonal antibody
* treatment with anti-TNF-α, methotrexate, cyclophosphamide, dapsone, methylprednisolone pulses or any other immunosuppressive or immunomodulatory drug or biotherapy within 6 months before inclusion
* long-course systemic GC therapy
* prednisone therapy >1 mg/kg/day, whatever the duration
* serious or chronic proven infections requiring hospitalization or intravenous antibiotics within 30 days before inclusion
* other proven infections that required antibiotics within 14 days before inclusion
* opportunistic infections
* evidence of active tuberculosis or latent tuberculosis (as deﬁned by a positive interferon gamma release assay)
* active chronic hepatitis B or C or HIV
* cancer or lymphoproliferative disorders within the 5 years before inclusion (with the exception of in situ cervical cancer and squamous or basal cell carcinoma with R0 resection)
* past history of sigmoid diverticulitis
* any active hepatic disease
* hepatic failure; thrombocytopenia <50 G/L
* neutropenia <0.5 G/L
* history of moderate to severe congestive heart failure or demyelinating disease
* recent stroke
* current signs or symptoms of severe, progressive, or uncontrolled disease, not due to GCA, which contraindicates TCZ
* severe and uncontrolled hypercholesterolemia
* high cardiovascular risk (former cerebral or coronary vascular event, or vascular risk >20% at 10 years according to the Framingham risk score [24]); dementia; non-compliant patients
* patients under ward of court, tutelage or legal guardianship.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06-13 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in remission with a dose of prednisone ≤ 0.1 mg/kg/day | Week 26
  Remission: absence of symptoms attributable to Giant Cell Arteritis and normalization of inflammatory markers (CRP<10 mg/L and ESR<30 mm/h).
  Relapse: recurrence of symptoms attributable to active GCA and/or increased levels of inflammatory markers (CRP≥10 mg/L and/or ESR≥30 mm/h). Elevation of inflammatory markers in the absence of GCA symptoms was considered relapse if it persisted at two time points at 1 week apart without any other obvious etiology than GCA.

SECONDARY OUTCOMES:
Frequency and type of adverse effects encountered | Until Week 52
Percentage of relapses | Week 26 and Week 52
Time to the first relapse | Until Week 52
Factors associated with the occurrence of relapse | Until Week 52
The cumulative dose of prednisone. | Weeks 26 and 52

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU de Caen - Hôpital Côte de Nacre, Caen
  - CHU de Dijon, Dijon
  - Chu Dupuytren, Limoges
  - Hôpital Edouard HERRIOT, Lyon
  - Hôpitaux privés de Metz - Site Sainte Blandine, Metz
  - Institut Mutualiste Montsouris, Paris
  - Hôpital La Pitié-Salpêtrière, Paris
  - Hôpital COCHIN, Paris

REFERENCES:
- [Derived] Samson M, Devilliers H, Ly KH, Maurier F, Bienvenu B, Terrier B, Charles P, Guillevin L, Besancenot JF, Liozon E, Fauchais AL, Loffroy R, Binquet C, Audia S, Seror R, Mariette X, Bonnotte B. Tocilizumab as an add-on therapy to glucocorticoids during the first 3 months of treatment of Giant cell arteritis: A prospective study. Eur J Intern Med. 2018 Nov;57:96-104. doi: 10.1016/j.ejim.2018.06.008. Epub 2018 Jul 24. PMID 30054122